CLINICAL TRIAL: NCT04924868
Title: Ursodeoxycolic Acid for the Prevention of Relapsing Complications After Gallstone Acute Pancreatitis, a Double-blind Multicenter Randomized-controlled Trial. OSOPOLAR Trial
Brief Title: Ursodeoxycolic Acid for the Prevention of Relapsing Complications After Gallstone Acute Pancreatitis
Acronym: OSOPOLAR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario de Alicante (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Enrique de-Madaria, Coordinator of Biliary-Pancreatic Unit., Hospital General Universitario de Alicante
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020/159; 2020-005901-16 (EudraCT Number)
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Acute Pancreatitis Due to Gallstones
Keywords: Acute pancreatitis; Gallstones; Ursodeoxycholic Acid; Randomized Controlled Trial
MeSH Terms: conditions — Pancreatitis; Gallstones | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UDCA (Ursodeoxycholic Acid) group (Active Comparator): Patients receiving Ursodeoxycholic Acid, capsules containing 300 mg, 10 mg/Kg per day:
  Patients 40 to 70 kg: 2 capsules/day >70 to 100 Kg: 3 capsules/day >100 kg: 4 capsules/day
  Interventions: Drug: Ursodeoxycholic Acid
- Placebo group (Placebo Comparator): Capsules containing placebo, indistinguishable from active treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — Ursodeoxycholic Acid will be administered to patients in the UDCA group as a prophylactic measure of future complications associated to gallstones
  Arms: UDCA (Ursodeoxycholic Acid) group
Drug: Placebo — Placebo: composition per 100g: colloidal silica 1.95g and cellulose microcrystalline 98.05g.
  Arms: Placebo group

SUMMARY:
Acute pancreatitis is a common disease (3rd cause of hospital admission for digestive causes), which is associated with significant patient suffering, a 2-4% probability of death and considerable healthcare costs. Sixty percent of acute pancreatitis are due to the presence of stones in the gallbladder. The risk of suffering another acute biliary pancreatitis (ABP, that is to say, pancreatitis due to gallstones) or of other biliary complications in the following weeks or months is high (20% or greater) if measures are not taken to avoid it, being surgical removal of the gallbladder the most effective. Unfortunately, most Spanish centers have a surgical waiting list that makes gallbladder surgery unfeasible in a period of less than weeks or months, which is why readmission for biliary problems derived from the stones is a common problem. This, of course, causes danger and great stress and anger for patients affected by these complications on the waiting list, damaging their relationship with the health system and it is linked to increased cost. In addition, there is a very vulnerable group, those patients who due to age or serious diseases cannot undergo gallbladder surgery but have a high probability of suffering biliary problems due to the stones they have.

Ursodeoxycholic acid (UDCA) is very safe drug which is used to dissolve gallstones, but its role in preventing biliary complications after ABP has not been studied adequately so it is not frequently used. Our objective is to investigate if UDCA is useful in this scenario, which would avoid suffering and adverse consequences for the patient and reduce the consumption of resources.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Hospital admission due to acute pancreatitis (definition: at least 2 of the following criteria: A) Typical pancreatitis pain, B) Amylase and/or lipase higher than 3 times the upper level of normality, C) Imaging compatible with acute pancreatitis
* Presence of gallstones according to any imaging technique
* Patient informed consent

Exclusion Criteria:

* Cholecystectomy and/or endoscopic retrograde cholangio-pancreatography and / or endoscopic cholecystostomy prior to recruitment
* Recurrent acute pancreatitis (1 or more previous episodes of pancreatitis of any origin)
* Current waiting list for cholecystectomy for acute biliary pancreatitis at that center less than 30 days
* Randomization more than 3 days after hospital discharge for acute pancreatitis
* Ursodeoxycholic acid (UDCA) consumption in the last 5 years or previous UDCA failure to dissolve lithiasis
* Allergy, intolerance or presence of contraindications to UDCA (contraindicated in patients with active gastric or duodenal ulcer, liver or intestinal disorders that interfere with the enterohepatic circulation of bile salts and lactation)
* Presence of choledocholithiasis diagnosed by imaging tests prior to randomization
* Active alcoholism greater than or equal to 5 daily alcoholic drinks in men or 3 in women or high clinical suspicion of clinically significant alcoholism
* Recent history of significant therapeutic non-compliance or social problem that makes follow-up difficult
* Hypertriglyceridemia greater than 400 mg / dL during admission or history of poorly controlled severe hypertriglyceridemia
* Chronic pancreatitis (pancreatic calcifications and / or Wirsung duct 4 or more mm)
* Pancreatic cystic lesions not attributed to the pancreatitis itself
* Wirsung duct stenosis
* Primary hyperparathyroidism
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Complication due to gallstones | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Composite endpoint: incidence of any of the following: acute pancreatitis, acute cholangitis, acute cholecystitis, biliary colic (with or without choledocholithiasis) Definitions are provided in "Secondary Outcome Measures"

SECONDARY OUTCOMES:
Relapse of acute pancreatitis | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  New episode of acute pancreatitis after recruitment Definition of acute pancreatitis (revised Atlanta classification): 2 or more of the following criteria: A) Typical pancreatitis pain, B) Amylase and/or lipase higher than 3 times the upper level of normality, C) Imaging compatible with acute pancreatitis
Incidence of acute cholangitis | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Acute cholangitis after recruitment
  Acute cholangitis definition (Tokyo 2018 guidelines):
  A. Systemic inflammation: A-1. Fever and/or shaking chills; A-2. Laboratory data: evidence of inflammatory response B. Cholestasis: B-1. Jaundice; B-2. Laboratory data: abnormal liver function tests C. Imaging: C-1. Biliary dilatation; C-2. Evidence of the etiology on imaging (stricture, stone, stent etc.) Suspected diagnosis: one item in A + one item in either B or C Definite diagnosis: one item in A, one item in B and one item in C
Incidence of acute cholecystitis | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Acute cholecystitis after recruitment
  Acute cholecystitis definition (Tokyo 2018 guidelines):
  A. Local signs of inflammation: (1) Murphy's sign, (2) RUQ mass/pain/tenderness B. Systemic signs of inflammation: (1) Fever, (2) elevated CRP, (3) elevated WBC count C. Imaging findings: Imaging findings characteristic of acute cholecystitis Suspected diagnosis: one item in A + one item in B Definite diagnosis: one item in A + one item in B + C
Incidence of biliary colic, with or without choledocholithiasis | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Biliary colic after recruitment Biliary colic definition: typical biliary colic pain. Choledocholithiasis: presence of stones or biliary sludge in the common bile duct according to imaging or endoscopic retrograde cholangio-pancreatography
Effectiveness of ursodeoxycholic acid in treating gallstones | Abdominal ultrasonography will be performed at 6 and 12 months after recruitment unless cholecystectomy is performed
  Decrease or elimination of gallstones according to ultrasonography
EORTC-QLQ C30 questionnaire | Measurement at 1, 3, 6, 9 and 12 months after recruitment
  EORTC-QLQ C30 questionnaire as a measure of Quality of Life
Hospital stay during follow-up | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Number of days admitted due to symptomatic gallstone disease
Intensive care unit stay during follow-up | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Number of days admitted in the intensive care unit due to symptomatic gallstone disease
Adverse events | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Adverse events due to ursodeoxycolic acid or placebo
Number of visits to emergency room or hospital admissions due to symptomatic gallstone disease | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Number of visits to emergency room or hospital admissions due to symptomatic gallstone disease
Need for endoscopic retrograde cholangio-pancreatography (ERCP) during follow-up | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Need for ERCP due to choledocholithiasis or acute cholangitis
Need for gallbladder endoscopic or percutaneous drainage during follow-up | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Need for gallbladder endoscopic or percutaneous drainage due to acute cholecystitis or cholangitis
Need for drainage of collections and abscesses | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Need for drainage of collections and abscesses (liver abscess, symtomatic pancreatic or peripancreatic collections not related to the index acute pancreatitis)
Incidence of organ failure during follow-up | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Organ failure definition (revised Atlanta classification): PaO2/FIO2<300, Creatinine >=1.9 mg/dl and/or systolic blood pressure <90mmHg despite fluid resuscitation
Mortality | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Death during follow-up
Need for urgent cholecystectomy | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Need for urgent cholecystectomy for acute gallbladder complication, mainly acute cholecystitis
Need for surgical necrosectomy | From recruitment to cholecystectomy or up to 1 year after recruitment if cholecystectomy is not performed
  Need for surgical necrosectomy, mainly after infection of pancreatic necrosis (not related to the index acute pancreatitis)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique De Madaria, Medicine, Principal Investigator — Alicante General University Hospital
Locations (18):
- Spain (18):
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A coruña
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Univerisitario Vall D´Hebron, Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Consorci Corporació Sanitària Parc Taulí de Sabadell, Sabadell, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Clínio San Cecilio, Granada, Granada
  - Hospital Ramon y Cajal, Madrid, Madrid
  - Hospital Costa del Sol,, Marbella, Málaga
  - Clinica Unversidad de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Ourense, Ourense, Ourense
  - Hospital Universitario Central de Asturias., Oviedo, Principality of Asturias
  - Hospital Clínico Universitario de Valencia, Alicante, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid
  - Hospital Universitario de Cruces, Bilbao, Vizcaya
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No